CLINICAL TRIAL: NCT03568838
Title: Prolonged Enoxaparin in Primary Percutaneous Coronary Intervention Compared With Standard of Care Therapy - The PENNYWISE Feasibility Study
Brief Title: Prolonged Enoxaparin in Primary Percutaneous Coronary Intervention
Acronym: PENNYWISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH19902
Record Dates: First submitted 2018-05-29; First posted 2018-06-26 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Patients will be randomised (1:1) using an opaque sealed envelope methodology prior to coronary angiography.
  Patients allocated to the experimental arm will receive a parenteral (IA/IV) bolus dose of enoxaparin (0.75 mg/kg) pre PPCI followed by an infusion of 0.75 mg/kg over a 6-hour period to be started as soon as possible when PPCI starts.
  Patients randomised to the standard therapy arm will receive treatment as guided by the treating cardiologist in line with the local standard-of-care, usually consisting of UFH and a GPI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin (Experimental): Patients allocated to the experimental arm will receive a parenteral (IA/IV) bolus dose of enoxaparin.
  Interventions: Drug: Enoxaparin
- Standard Therapy (No Intervention): Patients randomised to the standard therapy arm will receive treatment as guided by the treating cardiologist in line with the local standard-of-care, usually consisting of UFH and a GPI.

INTERVENTIONS:
Drug: Enoxaparin — Patients allocated to the experimental arm will receive a parenteral (IA/IV) bolus dose of enoxaparin (0.75 mg/kg) pre PPCI followed by an infusion of 0.75 mg/kg over a 6-hour period to be started as soon as possible when PPCI starts.
  Arms: Enoxaparin

SUMMARY:
This is a feasibility study aiming to generate pilot data on safety and efficacy of a novel anticoagulant regimen (enoxaparin bolus and prolonged infusion) compared to the local standard-of-care in opiate-treated patients undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Delayed absorption of oral P2Y12 inhibitors in patients undergoing primary percutaneous coronary intervention (PPCI) may increase the risk of stent thrombosis. Parenteral treatment is needed mitigate this risk.

We have recently shown a novel regimen of enoxaparin (bolus 0.75 mg/kg followed by an infusion of 0.75 mg/kg/6h) to provide consistent antithrombotic effects until the end of the infusion (1). We have also demonstrated the high prevalence of delayed platelet inhibition in opiate-treated patients (1).

This is a feasibility study for a larger randomised controlled trial (RCT). We aim to assess recruitment rate and collect pilot data on safety and efficacy. This will be a single-centre, open-label RCT comparing this novel regimen of enoxaparin to the local standard-of-care which usually consists of unfractionated heparin and a glycoprotein IIb/IIIa inhibitor. The study population will be opiate-treated patients undergoing PPCI. Pre PPCI, patients will be allocated in 1:1 ratio using a simple randomisation method using sealed envelopes, to either enoxaparin 0.75 mg/kg bolus followed by 0.75 mg/kg infusion over 6 hours (n=50) or the standard-of-care of UFH and tirofiban (n=50).

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Confirmation of the diagnosis of STEMI by the clinical team on the basis of history and ECG changes
* Intention to proceed with PPCI
* Treated with opiates for analgesia
* Feasibility to obtain informed verbal consent pre PPCI

Exclusion Criteria:

* Active bleeding that cannot be controlled by local measures
* Pregnant patients
* Patients with end-stage renal failure requiring renal replacement therapy
* Patients with cardiogenetic shock
* Known thrombocytopenia (Platelet count <100,000)
* Known history of intracranial haemorrhage
* Known current treatment with oral anticoagulants
* Known history of major surgery or trauma or history of GI/GU haemorrhage within the last month
* Known intracranial malignancy or aneurysm
* Known allergy to enoxaparin
* known hypersensitivity to benzylalcohol
* Patients with known acute bacterial endocarditis
* Known active gastric or duodenal ulceration
* Inability to easily understand verbal information given in English for any reason
* Inability to give informed consent due to either temporary or permanent mental incapacity
* Current participation, or participation within the last month, in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, average 1 year
  Recruitment rate over the study period
Bleeding rates within 24 hours | Through study completion, average 1 year
  These rates will be compared between the two treatment groups. Trivial bleeding related to access site will be excluded. Details on bleeding events will be collected and subsequently classified according to BARC types 2-5

SECONDARY OUTCOMES:
Acute stent thrombosis rate in each treatment arm | Through study completion, average 1 year
  Acute stent thrombosis rate in each treatment arm (within 24 hours). These rates will be compared between the two treatment groups.
Rates of ST-segment resolution in each treatment arm | Through study completion, average 1 year
  Comparison will be undertaken between presentation ECG and ECG performed 1 hour post PPCI. We will compare rates of ST segment resolution between the two treatment groups.
Rates of the composite outcomes | Through study completion, average 1 year
  Rates of the composite outcome of recurrent myocardial infarction, ischaemic stroke or cardiovascular death within 30 days of STEMI. These rates will be compared between the two treatment groups.
1-year mortality rates | Through study completion, average 1 year
  These will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Storey, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Sumaya W, Parker WAE, Fretwell R, Hall IR, Barmby DS, Richardson JD, Iqbal J, Adam Z, Morgan KP, Gunn JP, Mason AE, Judge HM, Gale CP, Ajjan RA, Storey RF. Pharmacodynamic Effects of a 6-Hour Regimen of Enoxaparin in Patients Undergoing Primary Percutaneous Coronary Intervention (PENNY PCI Study). Thromb Haemost. 2018 Jul;118(7):1250-1256. doi: 10.1055/s-0038-1657768. Epub 2018 Jun 6. PMID 29874689